CLINICAL TRIAL: NCT00262782
Title: Prognostic Factors and Risk-Adapted Therapy in Patients With Early Stage Chronic Lymphocytic Leukemia
Brief Title: Fludarabine or Observation in Treating Patients With Stage 0, Stage I, or Stage II Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL1; EU-20548; GCLLSG-138; MEDAC-GCLLSG-CLL1
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine

ARMS (2):
- Fludarabine (Experimental)
  Interventions: Drug: Fludarabine
- watch & wait (No Intervention)

INTERVENTIONS:
Drug: Fludarabine — Fludarabine i.v. (25 mg/m2/d, d1-5) q28d; max 6 cycles
  Other Names: Fludura
  Arms: Fludarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Sometimes, the cancer may not need treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether fludarabine is more effective than observation in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying fludarabine to see how well it works compared to observation only in treating patients with stage 0, stage I, or stage II B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify prognostic factors that predict a short survival in patients with stage 0-II B-cell chronic lymphocytic leukemia treated with fludarabine or observation only.

OUTLINE: This is a randomized study. Patients are stratified according to risk (high risk vs low risk). Patients in the low-risk group undergo observation only. Patients in the high-risk group are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine.
* Arm II: Patients undergo observation only.

PROJECTED ACCRUAL: A total of 880 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of B-cell chronic lymphocytic leukemia

  * Rai stage 0-II (Binet stage A) disease
* Meets 1 of the following criteria:

  * High-risk disease, as defined by the following:

    * Serum thymidine kinase level > 7.0 U/L
    * Elevated β2-microglobulin level
    * Presence of non-nodular bone marrow infiltration
    * Short lymphocyte doubling time
  * Low-risk disease

    * Meets none of the criteria (as listed above) for high-risk disease

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* More than 6 months

Hematopoietic

* No autoimmune hemolytic anemia
* No thrombocytopenia

Hepatic

* Not specified

Renal

* Not specified

Other

* No severe organ dysfunction
* No other prior or concurrent malignancy

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 1997-04; Primary Completion 2004-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (115):
- Austria (2):
  - Allg. Krankenhaus der Stadt Wien Universitaets-Kinderklinik, Vienna
  - Hanuschkrankenhaus, Vienna
- Germany (113):
  - Klinikum St. Marien, Amberg
  - Internistische Praxis - Arnstadt, Arnstadt
  - Zentralklinikum Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Regional Hospital Am Plattenwald, Bad Friedrichshall
  - Regional Hospital Bad Hersfeld, Bad Hersfeld
  - Arzt fuer Innere Medizin - Bad Reichenhall, Bad Reichenhall
  - Humaine - Clinic, Bad Saarow
  - Ermstalklinik Bad Urach, Bad Urach
  - Internistische Praxis - Berlin, Berlin
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Haematologisch-Onkologische Schwerpunktpraxis, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite - Campus Virchow Klinikum, Berlin
  - Gemeinschaftspraxis - Betzdorf, Betzdorf
  - Praxis Dres. F.& G. Doering, Bremen
  - Krankenhaus Burglengenfeld, Burglengenfeld
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Onkologische Schwerpunktpraxis, Cottbus
  - Staedtisches Klinikum Dessau, Dessau
  - Onkologische Gemeinschaftspraxis - Dresden, Dresden
  - Michael Schaefers und Partner, Duisburg
  - Universitaetsklinik Duesseldorf, Düsseldorf
  - Internistische Gemeinschaftpraxis - Ehingen, Ehingen
  - Onkologische Schwerpunktpraxis - Erding, Erding
  - Internistische/Onkologische Praxis - Erfurt, Erfurt
  - Onkologische Schwerpunkt Praxis, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Internistische Gemeinschaftspraxis - Forchheim, Forchheim
  - Klinikum Garmisch - Partenkirchen, Garmisch-Partenkirchen
  - Gemeinschaftspraxis - Germering, Germering
  - Internistische Praxisgemeinschaft, Germering
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Onkologische Gemeinschaftspraxis - Gross-Gerau, Groß-Gerau
  - St. Marien Hospital at Katholisches Krankenhaus hagen gem. GmbH, Hagen
  - Allgemeines Krankenhaus Hagen, Hagen
  - Internistische Praxis - Halle, Halle
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - Martin Luther Universitaet, Halle
  - Praxis fur Innere Medizin - Hamburg, Hamburg
  - Allgemeines Krankenhaus St. Georg, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Schwerpunktpraxis Haematologie/Onkologie - Hannover, Hanover
  - Facharzt fuer Allgemeinmedizin - Hausham, Hausham
  - Facharzt fuer Innere Medizin - Hechingen, Hechingen
  - Onkologische Schwerpunktpraxis Heidelberg, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Medizinischen Klinik Dr. R. Schindlbeck, Herrsching am Ammersee
  - Oncological Specialist Practice, Hildesheim
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Praxis am Evangelischen Krankenhaus Bethanien, Iserlohn
  - Internistische Gemeinschaftspraxis - Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Staedt Klinikum Karlsruhe GGMBH, Karlsruhe
  - Facharzt Fuer Jnnere Medizin, Karlsruhe
  - St. Vincentius-Kliniken, Karlsruhe
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Staedtische Krankenhaus Kiel, Kiel
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Onkologische Schwerpunktpraxis Leer, Leer
  - Klinikum Lippe - Lemgo, Lemgo
  - Universitaetsklinkum Magdeburg der Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
  - Gemeinschaftspraxis, Mannheim
  - Philipps-Universitaet Marburg Klinikum, Marburg
  - Internistische Gemeinschaftspraxis - Memmingen, Memmingen
  - Klinikum Minden, Minden
  - Haematologische Praxis - Moenchengladbach, Mönchengladbach
  - Klinikum Innenstadt, Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Hamatologische Schwerpunktpraxis, Munich
  - Munich Oncologic Practice at Elisenhof, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinikum Garmisch-Partenkirchen GmbH Abteilung fuer Innere Medizin Murnau, Murnau am Staffelsee
  - Haematologisch-onkologische Gemeinschaftspraxis - Muenster, Münster
  - Internistische Praxis - Neuenkirchen, Neuenkirchen
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Sudharz-Krankenhaus Nordhausen gGmbH, Nordhausen
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Hematologische Praxis, Oldenburg
  - Gemeinschaftliche Schwerpunktpraxis - Osnabrueck, Osnabrück
  - Municipal Hospital Complex, Pforzheim
  - Hematologische Onkologische Praxis, Regensburg
  - Jakobi Krankenhaus, Rheine
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Schwerpunktpraxis Fuer Haematologie Und Onkologie, Saarbruecke
  - Caritasklinik St. Theresia, Saarbrücken
  - Onkologische Schwerpunktpraxis - Schrobenhausen, Schrobenhausen
  - Praxis - Schwenningen, Schwenningen
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Evang. Jung-Stilling Hospital, Siegen
  - Praxisgemeinschaft - Stade, Stade
  - Onkologische Schwerpunktpraxis - Straubing, Straubing
  - Haematologische Praxis, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Onkologische Gemeinschaftspraxis - Trier, Trier
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - St. Marien Hospital, Vechta
  - Gemeinschaftspraxis - Weiden, Weiden
  - Haematologisch-Onkologische Schwerpunktpraxis - Weilheim, Weilheim
  - Internistische Praxis - Wendlingen, Wendlingen
  - Kliniken St. Antonius, Wuppertal
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg
  - Medizinische Klinik und Poliklinik II - Universitaetsklinikum Wuerzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gobel M, Eisele L, Mollmann M, Huttmann A, Johansson P, Scholtysik R, Bergmann M, Busch R, Dohner H, Hallek M, Seiler T, Stilgenbauer S, Klein-Hitpass L, Duhrsen U, Durig J. Progranulin is a novel independent predictor of disease progression and overall survival in chronic lymphocytic leukemia. PLoS One. 2013 Aug 23;8(8):e72107. doi: 10.1371/journal.pone.0072107. eCollection 2013. PMID 24009671
- [Background] Sachanas S, Pangalis GA, Fink AM, Bahlo J, Fischer K, Levidou G, Kyrtsonis MC, Bartzi V, Vassilakopoulos TP, Kalpadakis C, Koulieris E, Moschogiannis M, Yiakoumis X, Tsirkinidis P, Angelopoulou MK, Eichhorst B, Hallek M. Small Lymphocytic Lymphoma: Analysis of Two Cohorts Including Patients in Clinical Trials of the German Chronic Lymphocytic Leukemia Study Group (GCLLSG) or in "Real-Life" Outside of Clinical Trials. Anticancer Res. 2019 May;39(5):2591-2598. doi: 10.21873/anticanres.13382. PMID 31092457
- [Result] Bergmann MA, Eichhorst BF, Busch R, et al.: Early and risk-adapted therapy with fludarabine in high-risk Binet stage A CLL patients prolongs progression free survival but not overall survival: results of the CLL1 protocol of the German CLL Study Group (GCLLSG). [Abstract] Blood 110 (11): A-2038, 2007.
- [Result] Bergmann MA, Eichhorst BF, Busch R, et al.: Prospective evaluation of prognostic parameters in early stage chronic lymphocytic leukemia (CLL): results of the CLL1-protocol of the German CLL Study Group (GCLLSG). [Abstract] Blood 110 (11): A-625, 2007.
- [Result] Hoechstetter MA, Busch R, Eichhorst B, Buhler A, Winkler D, Eckart MJ, Vehling-Kaiser U, Schimke H, Jager U, Hurtz HJ, Hopfinger G, Hartmann F, Fuss H, Abenhardt W, Blau I, Freier W, Muller L, Goebeler M, Wendtner CM, Bahlo J, Fischer K, Bentz M, Emmerich B, Dohner H, Hallek M, Stilgenbauer S. Early, risk-adapted treatment with fludarabine in Binet stage A chronic lymphocytic leukemia patients: results of the CLL1 trial of the German CLL study group. Leukemia. 2017 Dec;31(12):2833-2837. doi: 10.1038/leu.2017.246. Epub 2017 Aug 14. No abstract available. PMID 28804126
- [Result] Hoechstetter MA, Busch R, Eichhorst B, Buhler A, Winkler D, Bahlo J, Robrecht S, Eckart MJ, Vehling-Kaiser U, Jacobs G, Jager U, Hurtz HJ, Hopfinger G, Hartmann F, Fuss H, Abenhardt W, Blau I, Freier W, Muller L, Goebeler M, Wendtner C, Fischer K, Herling CD, Starck M, Bentz M, Emmerich B, Dohner H, Stilgenbauer S, Hallek M. Prognostic model for newly diagnosed CLL patients in Binet stage A: results of the multicenter, prospective CLL1 trial of the German CLL study group. Leukemia. 2020 Apr;34(4):1038-1051. doi: 10.1038/s41375-020-0727-y. Epub 2020 Feb 10. PMID 32042081
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Jaramillo S, Agathangelidis A, Schneider C, Bahlo J, Robrecht S, Tausch E, Bloehdorn J, Hoechstetter M, Fischer K, Eichhorst B, Goede V, Hallek M, Dohner H, Rosenquist R, Ghia P, Stamatopoulos K, Stilgenbauer S. Prognostic impact of prevalent chronic lymphocytic leukemia stereotyped subsets: analysis within prospective clinical trials of the German CLL Study Group (GCLLSG). Haematologica. 2020 Nov 1;105(11):2598-2607. doi: 10.3324/haematol.2019.231027. PMID 33131249
- [Derived] Kreuzberger N, Damen JA, Trivella M, Estcourt LJ, Aldin A, Umlauff L, Vazquez-Montes MD, Wolff R, Moons KG, Monsef I, Foroutan F, Kreuzer KA, Skoetz N. Prognostic models for newly-diagnosed chronic lymphocytic leukaemia in adults: a systematic review and meta-analysis. Cochrane Database Syst Rev. 2020 Jul 31;7(7):CD012022. doi: 10.1002/14651858.CD012022.pub2. PMID 32735048
- [Derived] Pflug N, Bahlo J, Shanafelt TD, Eichhorst BF, Bergmann MA, Elter T, Bauer K, Malchau G, Rabe KG, Stilgenbauer S, Dohner H, Jager U, Eckart MJ, Hopfinger G, Busch R, Fink AM, Wendtner CM, Fischer K, Kay NE, Hallek M. Development of a comprehensive prognostic index for patients with chronic lymphocytic leukemia. Blood. 2014 Jul 3;124(1):49-62. doi: 10.1182/blood-2014-02-556399. Epub 2014 May 5. PMID 24797299